CLINICAL TRIAL: NCT02696486
Title: Exercise Training Effect on Quality of Life and Exercise Capacity in Patients With Heart Failure and Preserved Ejection Fraction: A Pilot Study
Brief Title: Exercise Training Effect in Patients With HF and PEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MultiCare Health System Research Institute (Other)
Collaborators: Henry Ford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15.20
Record Dates: First submitted 2016-02-22; First posted 2016-03-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Training (Experimental)
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training — Study subjects will receive medically supervised aerobic and resistance exercise training for 1 hour per session, 3 times per week for 6 weeks at the Cardiac Rehab center and then transition to home or YMCA partnership based exercise with staff follow-up contact for an additional 3 weeks.

SUMMARY:
The purpose of this is to develop and implement a pilot study that will demonstrate the ability to recruit, enroll, retain, conduct exercise training, and collect pre and post outcomes on the effect of exercise training on quality of life (QOL) and exercise capacity in patients with a diagnosis of heart failure with preserved ejection fraction (HFPEF).

ELIGIBILITY:
Inclusion Criteria:

* Age > 55 years (Interested in capturing mean ages close to age 65 as many HF initiatives are based on this age group and HF development increases with aging).
* Diagnosis of HFPEF stable NYHA Stage II- III with an EF of ≥ 45%
* Stabilized on cardiac medications and post hospitalization > 4 weeks
* Ability to participate in exercise testing and training.
* Referral from Cardiologist or primary care physician.

Exclusion Criteria:

* Unstable Angina
* Uncontrolled diabetes
* Moderate to severe aortic stenosis
* Uncontrolled hypertension Systolic BP>150 mm Hg or Diastolic BP >100 mm Hg
* Valvular heart disease
* Untreated coronary artery stenosis >50%
* Arrhythmias
* Pulmonary disease/COPD
* Dementia or cognitive impairment
* VAD or Transplant planned in next 6 months.
* Current or recent participation in a Cardiac Rehab program within the last six months.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11; Primary Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life (QOL) score pre and post exercise training (ET). | 9 weeks

SECONDARY OUTCOMES:
Change in exercise capacity/tolerance pre and post ET using Cardiopulmonary Exercise Testing. | 9 weeks
  Symptom limited treadmill testing with expired gas measurement and analysis. Exercise capacity measured as Peak Vo2 (peak exercise oxygen uptake) in ml/min/kg. Continuous monitoring of 12 lead electrocardiogram and blood pressure measured every 2 minutes. Peak Vo2 defined as highest Vo2 value of the last 30 seconds before termination of exercise. Exercise time and peak workload will be measured for exercise tolerance.
Demonstrated ability to coordinate patient transition from clinic to home or YMCA partnership based exercise program with weekly staff follow-up within the study timeline. | 9 weeks
Capture 90 day hospital readmission data starting with study enrollment date and within the participants' study timeline. | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- MultiCare Health System, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bean G, Mou J, Pflugeisen B, Olsen L, Hoag S, Silva A, Ball AL, Lee T. Exercise Training in Patients With Heart Failure With Preserved Ejection Fraction: A Community Hospital Pilot Study. J Cardiovasc Nurs. 2021 Mar-Apr 01;36(2):124-130. doi: 10.1097/JCN.0000000000000737. PMID 32740221